CLINICAL TRIAL: NCT07125066
Title: An Individual Patient, Open Label Study to Use ACER-001 to Treat Combined D,L-2-hydroxyglutaric Aciduria (C-2HGA)
Brief Title: An Individual Patient, Open Label Study to Use ACER-001 to Treat Combined D,L-2 Hydroxyglutaric Aciduria (C-2HGA)
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Jerry Vockley, MD, PhD (Other)
Collaborators: Zevra Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Jerry Vockley, MD, PhD, Chief, Division of Genetic and Genomic Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25060137
Record Dates: First submitted 2025-07-30; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Combined D,L-2-hydroxyglutaric Aciduria
Keywords: Combined D,L-2-hydroxyglutaric aciduria
MeSH Terms: interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- sodium phenylbutyrate (Experimental): a single patient will take sodium phenylbutyrate (ACER-001) current at a dose of 12 g/day; dose will be modified if the patient gains more than 5 kg of weight
  Interventions: Drug: Sodium phenylbutyrate

INTERVENTIONS:
Drug: Sodium phenylbutyrate — open-label design with doses of sodium phenylbutyrate
  Other Names: Olpruva

SUMMARY:
This is an individual patient research protocol to treat a patient diagnosed with Combined D,L-2-hydroxyglutaric aciduria (C-2HGA) with ACER-001.

DETAILED DESCRIPTION:
Patient will continue to be seen during routine outpatient clinic visits every 6 months. At those visits the following will be collected: routine metabolic laboratory tests (including a complete metabolic profile, complete blood count, blood phenylacetylglutamine level, and urine organic acids), physical examinations, and an update of clinical history, especially regarding seizures and respiratory status.

Once consent is signed, the patient will continue to take ACER-001 as prescribed. The ACER-001 will be provided to the patient at no cost.

ELIGIBILITY:
Inclusion Criteria:

* Single patient with Combined D,L-2-hydroxyglutaric aciduria
* Parental permission must be given at the start of the protocol.
* Parents willing to adhere to the protocol

Exclusion Criteria:

* Refusal or withdrawal of consent.
* Drug Intolerance.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of treatment related adverse events | 2 years

SECONDARY OUTCOMES:
Change in the amount of urine D,L 2-Hydroxyglutaric acid in urine | 2 years
Change in phenylacetylglutamine in urine | 2 years
Change in the number of seizures reported by parents | 2 years
Change in ventilator support | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Vockley, MD, PhD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No